CLINICAL TRIAL: NCT04283123
Title: Evaluating the Feasibility of an Automated Bidet Intervention to Decrease Caregiver Burden
Brief Title: Feasibility of an Automated Bidet Intervention to Decrease Caregiver Burden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Susan Stark, Associate Professor of Occupational Therapy, Neurology and Social Work, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201610044
Record Dates: First submitted 2020-02-14; First posted 2020-02-25 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Caregiver Burnout
Keywords: Assistive Technology; Informal Caregivers; Occupational Therapy; Toileting
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants assigned to this group will receive an automated bidet (TOTO Washlet S300e with remote control) and an occupational therapy intervention over 2-3 in-home visits.
  Interventions: Behavioral: Automated Bidet
- Waitlist Control (Active Comparator): Caregivers will wait for 30 days and then will be offered the intervention.
  Interventions: Other: No Intervention

INTERVENTIONS:
Behavioral: Automated Bidet — During the first intervention visit, a licensed contractor will install the bidets in participants' homes. The OT will then educate and train the caregiver and care recipient to successfully use the bidet, and make any modifications to the remote as needed. Throughout the intervention, the OT will use motivational enhancement strategies. The OT will make minor modifications to the remote as needed. A second intervention visit will occur 1-2 weeks post-installation to address any new difficulties. Check-in phone calls will be offered to the caregiver and care recipient if needed.
  Arms: Treatment
Other: No Intervention — Waitlist control
  Arms: Waitlist Control

SUMMARY:
This study evaluates the feasibility, including acceptability and preliminary efficacy, of an automated bidet intervention to make it easier for caregivers to assist with toileting.

DETAILED DESCRIPTION:
Informal caregivers provide over 30 billion hours of care to older adults each year. They often assist with toileting tasks which are often identified as one of the most physically and emotionally demanding activities of daily living. Caregivers receive limited training and support which increases their risk for injury and burnout. One potential strategy to reduce or replace the physical support needed from a caregiver is the used of an automated bidet system. It remains unknown whether an automated bidet can be used successfully with older adults and their caregivers at home. The objective of this feasibility study was to assess the acceptability and preliminary efficacy of a toileting intervention using an automated bidet system and training by an occupational therapy practitioner (OT) to reduce the amount of physical assistance required from caregivers.

The investigators will recruit 10 informal caregivers and randomize them to the treatment or waitlist control group. Caregivers in the treatment group will receive the automated bidet right away while those in the waitlist control group will not receive any treatment during that time. After 30 days, both groups will participate in a post-test assessment visit. The waitlist control group will then be offered the intervention and invited to participate in a final session after 30 days to complete assessments and a process evaluation (30 days post follow-up).

ELIGIBILITY:
Inclusion Criteria:

* (1) provided unpaid care and lived with a care recipient aged 55 years or older
* (2) assisted with toileting for at least 6 months
* (3) did not have an automated bidet
* (4) had a working toilet and bathroom outlet, and (5) their care recipient was willing to participate

Exclusion Criteria:

* Caregivers scoring 10 or above on the Short Blessed Test, indicating possible cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stark, PhD, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We contacted 55 informal caregivers from December 2016 to April 2017. Twenty-four(43.6%) expressed interest in participating, but 14 were ineligible (7 did not provide toileting assistance; 3 primarily used a commode or absorbent underwear; 2 had paid caregivers; 1did not meet the age criterion; and 1 care recipient was interested, but the caregiver was not). Ten informal caregivers were enrolled in this study.
Groups:
- Treatment: Participants assigned to this group will receive an automated bidet (TOTO Washlet S300e with remote control) and an occupational therapy intervention over 3-4 in-home visits.
  Automated Bidet: During the first intervention visit, a licensed contractor will install the bidets in participants' homes. The OT will then educate and train the caregiver and care recipient to successfully use the bidet, and make any modifications to the remote as needed. Throughout the intervention, the OT will use motivational enhancement strategies. The OT will make minor modifications to the remote as needed. A second intervention visit will occur 1-2 weeks post-installation to address any new difficulties. Check-in phone calls will be offered to the caregiver and care recipient if needed.
Period: Overall Study
Arm/Group | Treatment | Waitlist Control
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Waitlist Control | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.40 (10.29) | 64.40 (14.19) | 66.40 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited
Description: The ability to recruit 10 caregivers who were eligible for the study was used with other variables to assess feasibility
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Waitlist Control
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

2. Primary Outcome: Number of Caregivers Retained
Description: Retain 10 caregivers was used with other variables to assess feasibility
Time Frame: At study completion (2 months [treatment] or 3 months [waitlist control])
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Waitlist Control
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

3. Primary Outcome: Number of Participants With Ability to Install the Automated Bidets, Including Any Modifications Needed
Description: Installation of the automated bidets and a record of any modifications needed was used with other variables to assess feasibility
Time Frame: 30 days post-installation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Waitlist Control
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

4. Primary Outcome: Number of Caregivers' or Care Recipients' Who Can Operate the Bidet
Description: Demonstrate ability to operate the bidet successfully which was used with other variables to assess feasibility
Time Frame: 30 days post-installation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Waitlist Control
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

5. Primary Outcome: Acceptability
Description: 8-item process evaluation: rated on a scale of 0 (strongly disagree) to 4 (strongly agree) with higher scores indicating greater acceptance of the intervention
Time Frame: 30 days post-installation
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total: All participants combined
Arm/Group | Treatment | Waitlist Control | Total
Number analyzed (Participants) | 5 | 5 | 10
units on a scale
  The automated bidet system was aesthetically pleasing/looked nice. | 3.60 (0.55) | 4.00 (0.00) | 3.80 (0.42)
  The automated bidet system was easy to use | 3.60 (0.55) | 4.00 (0.00) | 3.80 (0.42)
  The education and training on using the automated bidet system was very helpful | 4.00 (0.00) | 4.00 (0.00) | 4.00 (0.00)
  The automated bidet system made it easier for me to help my loved one with toileting | 3.80 (0.45) | 3.80 (0.45) | 3.80 (0.42)
  I feel more confident assisting my loved one with toileting tasks | 3.20 (0.84) | 3.80 (0.45) | 3.50 (0.71)
  The automated bidet addressed my concerns for providing assistance with toileting in the home | 3.20 (0.45) | 3.60 (0.55) | 3.40 (0.52)
  We will continue to use the automated bidet system after the conclusion of the study | 4.00 (0.00) | 4.00 (0.00) | 4.00 (0.00)
  The presence of my loved one during study visits impacted my ability to answer questions truthfully | 3.40 (1.34) | 4.00 (0.00) | 3.70 (0.95)

6. Primary Outcome: Preliminary Efficacy: Performance
Description: In-Home Occupational Performance Evaluation for Providing Assistance impact on caregiver outcomes rated on a scale of 1 to 5 with higher scores indicating better performance was used with other variables to assess feasibility
Time Frame: 2 months (treatment) or 3 months (waitlist control)
Population: The I-HOPE Assist was completed with caregivers at pretest and posttest (30 days post-intervention for the treatment group or 30 days post-enrollment for the control group), and at follow-up for the waitlist control group (30 days post-installation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Waitlist Control
Number analyzed (Participants) | 5 | 5
units on a scale
  Pretest | 3.20 (1.30) | 4.20 (0.84)
  Posttest | 4.20 (0.45) | 3.40 (0.89)
  Follow-up: number analyzed (Participants) | 0 | 5
  Follow-up |  | 4.40 (0.55)
Statistical Analysis 1: Comparison: Treatment; Test type: Other — Wilcoxon-signed rank test to compare differences from pretest to posttest for the treatment group. The standardized effect size was interpreted using Cohen's criteria; Cohen's d = 0.41 — Wilcoxon-signed rank test to compare differences from pretest to posttest for the treatment group. The standardized effect size was interpreted using Cohen's criteria
Statistical Analysis 2: Comparison: Waitlist Control; Test type: Other — Wilcoxon-signed rank test to compare differences from pretest to posttest for the waitlist control group. The standardized effect size was interpreted using Cohen's criteria; Cohen's d = 0.45 — Wilcoxon-signed rank test to compare differences from pretest to posttest for the waitlist control group. The standardized effect size was interpreted using Cohen's criteria

7. Primary Outcome: Preliminary Efficacy: Satisfaction
Description: In-Home Occupational Performance Evaluation for Providing Assistance: impact on caregiver outcomes rated on a scale of 1 to 5 with higher scores indicating better satisfaction was used with other variables to assess feasibility
Time Frame: 2 months (treatment) or 3 months (waitlist control)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Waitlist Control
Number analyzed (Participants) | 5 | 5
units on a scale
  Pretest | 3.20 (1.48) | 3.40 (1.14)
  Posttest | 4.40 (0.55) | 3.00 (0.71)
  Follow-up: number analyzed (Participants) | 0 | 5
  Follow-up |  | 4.60 (0.55)
Statistical Analysis 1: Comparison: Treatment; Test type: Other — [test comment as in outcome 6, analysis 1]; Cohen's d = 0.48 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Waitlist Control; Test type: Other — [test comment as in outcome 6, analysis 2]; Cohen's d = 0.32 — [estimate comment as in outcome 6, analysis 2]

8. Primary Outcome: Preliminary Efficacy: Self-efficacy
Description: In-Home Occupational Performance Evaluation for Providing Assistance: impact on caregiver outcomes rated on a scale of 1 to 5 with higher scores indicating better self-efficacy was used with other variables to assess feasibility
Time Frame: 2 months (treatment) or 3 months (waitlist control)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Waitlist Control
Number analyzed (Participants) | 5 | 5
units on a scale
  Pretest | 3.20 (1.30) | 3.60 (1.52)
  Posttest | 4.60 (0.55) | 3.60 (0.55)
  Follow-up: number analyzed (Participants) | 0 | 5
  Follow-up |  | 4.80 (0.45)
Statistical Analysis 1: Comparison: Treatment; Test type: Other — [test comment as in outcome 6, analysis 1]; Cohen's d = 0.60 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Waitlist Control; Test type: Other — [test comment as in outcome 6, analysis 2]; Cohen's d = 0.12 — [estimate comment as in outcome 6, analysis 2]

9. Primary Outcome: Preliminary Efficacy: Physical Environmental Barriers
Description: In-Home Occupational Performance Evaluation for Providing Assistance: reduction of physical barriers to toileting (rated on a scale from 0 (independent) to 5 (no activity/dependent) was used with other variables to assess feasibility
Time Frame: 2 months (treatment) or 3 months (waitlist control)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Waitlist Control | Total
Number analyzed (Participants) | 5 | 5 | 10
units on a scale
  Pretest | 10.20 (3.70) | 9.00 (3.39) | 9.60 (3.41)
  Posttest | 8.20 (3.11) | 8.60 (3.36) | 8.40 (3.06)
  Follow-up: number analyzed (Participants) | 0 | 5 | 5
  Follow-up |  | 6.40 (2.70) | 6.40 (2.70)

10. Primary Outcome: Adverse Events
Description: Number of adverse events was used with other variables to assess feasibility
Time Frame: At study completion (2 months [treatment] or 3 months [waitlist control])
Measure: Number; unit: adverse events
Arm/Group | Treatment | Waitlist Control
Number analyzed (Participants) | 5 | 5
adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to study completion (2 months [treatment] or 3 months [waitlist control])
Arm/Group | Treatment | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT04283123/Prot_SAP_000.pdf